CLINICAL TRIAL: NCT05045287
Title: Phase II Study of Hypofractionated Post Mastectomy Radiation With Two-Stage Expander/Implant Reconstruction
Brief Title: Hypofractionated Post Mastectomy Radiation With Two-Stage Expander/Implant Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jing Jin, M.D., Chief Physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS2021-6-1
Record Dates: First submitted 2021-08-24; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Breast Carcinoma
Keywords: hypofractionated radiotherapy; Two-Stage Expander/Implant Reconstruction; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hypofractionated radiation therapy (Experimental): receive chest wall and nodal irradiation at a dose of 43.5 Gy in 15 fractions over 3 weeks
  Interventions: Radiation: hypofractionated radiotherapy

INTERVENTIONS:
Radiation: hypofractionated radiotherapy — Undergo hypofractionated RT，obeserve reconstruction failure，cosmetic result and recurrence rate

SUMMARY:
Hypofractionated radiotherapy could provide more convenient treatment and had similar toxicities.However,reports of hypofractionated radiotherapy with two-stage expander/implant reconstruction are rare,Some studies have shown that hypofractionated radiotherapy had similar toxicities to conventional fractionated radiotherapy in patients with breast reconstruction. So,investigators conducted a phase II study to observe the reconstruction failure in hypofractionated radiotherapy with two-stage expander/implant reconstruction.

DETAILED DESCRIPTION:
Results from a phase III randomized controlled study in China showed that Postmastectomy hypofractionated radiotherapy was non-inferior to and had similar toxicities to conventional fractionated radiotherapy in patients with high-risk breast cancer.However,reports of hypofractionated radiotherapy with two-stage expander/implant reconstruction are rare. Literatures report that reconstruction failure is a well-known complication of radiation therapy in breast cancer patients with reconstruction. Results may vary based on RT timing and technique. Some studies have shown that hypofractionated radiotherapy had similar reconstruction failure to conventional fractionated radiotherapy in patients with breast reconstruction. So,investigators conducted a phase II study to observe the reconstruction failure in hypofractionated radiotherapy with two-stage expander/implant reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of stage I-IIIc invasive breast cancer (ductal, lobular, mammary, medullary, or ductal)

  ≤ T3 or N+
* negative surgery margins
* positive postoperative pathologic axillary lymph nodes after neoadjuvant chemotherapy (ypN+).
* Undergo mastectomy+expander+RT（hypofractionated radiotherapy）+delayed prosthesis reconstruction
* Sign the informed consent form

Exclusion Criteria:

* T4,
* axillary sentinel lymph node biopsy without axillary dissection
* Recurrent breast cancer or history of prior breast radiation therapy (neck, chest wall, axilla)
* Uncontrollable co-morbidities, including but not limited to active collagen vascular disease (e.g., systemic lupus erythematosus, scleroderma, or dermatomyositis), persistent or active infection, symptomatic congestive heart failure, unstable angina, mental illness incapacitating participation in this study
* Pregnancy or breastfeeding
* History of malignancy other than the following： (At least 5 years of tumor free survival with a very low risk of recurrence, e.g., carcinoma in situ of the cervix and basal cell or squamous cell carcinoma of the skin）
* requiring bilateral breast/chest wall radiation therapy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2021-04-08 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
reconstruction failure | 12 months after the reconstructive surgery
  the 1-year rate of implant removal due to serious complications (such as infection, hematoma, seromatas, prosthesis exposure, prosthesis rupture, envelope contracture, severe breast deformity, etc.)

SECONDARY OUTCOMES:
cosmetic result | 12 months after the reconstructive surgery
  Digital photographs will be taken of each patient to facilitate thorough assessment of breast symmetry, cleavage and donor site scarring. Overall satisfaction is scored on a five-point Likert scale (1 = very unhappy, 5 = very happy).

OTHER OUTCOMES:
Acute and late radiotherapy toxicity | through study completion, an average of 1 year
  Radiotherapy toxicity assessed by CTCAE3 and RTOG standard （e. g. acute skin toxicity, radiation pneumo nitis, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Jing jin, MD, Principal Investigator — Director of radiotherapy department
Locations (1):
- Jiawei Lu, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Khan AJ, Poppe MM, Goyal S, Kokeny KE, Kearney T, Kirstein L, Toppmeyer D, Moore DF, Chen C, Gaffney DK, Haffty BG. Hypofractionated Postmastectomy Radiation Therapy Is Safe and Effective: First Results From a Prospective Phase II Trial. J Clin Oncol. 2017 Jun 20;35(18):2037-2043. doi: 10.1200/JCO.2016.70.7158. Epub 2017 May 1. PMID 28459606
- [Result] Fowble B, Park C, Wang F, Peled A, Alvarado M, Ewing C, Esserman L, Foster R, Sbitany H, Hanlon A. Rates of Reconstruction Failure in Patients Undergoing Immediate Reconstruction With Tissue Expanders and/or Implants and Postmastectomy Radiation Therapy. Int J Radiat Oncol Biol Phys. 2015 Jul 1;92(3):634-41. doi: 10.1016/j.ijrobp.2015.02.031. Epub 2015 Apr 28. PMID 25936815
- [Result] Wang SL, Fang H, Song YW, Wang WH, Hu C, Liu YP, Jin J, Liu XF, Yu ZH, Ren H, Li N, Lu NN, Tang Y, Tang Y, Qi SN, Sun GY, Peng R, Li S, Chen B, Yang Y, Li YX. Hypofractionated versus conventional fractionated postmastectomy radiotherapy for patients with high-risk breast cancer: a randomised, non-inferiority, open-label, phase 3 trial. Lancet Oncol. 2019 Mar;20(3):352-360. doi: 10.1016/S1470-2045(18)30813-1. Epub 2019 Jan 30. PMID 30711522
- [Result] Santosa KB, Chen X, Qi J, Ballard TNS, Kim HM, Hamill JB, Bensenhaver JM, Pusic AL, Wilkins EG. Postmastectomy Radiation Therapy and Two-Stage Implant-Based Breast Reconstruction: Is There a Better Time to Irradiate? Plast Reconstr Surg. 2016 Oct;138(4):761-769. doi: 10.1097/PRS.0000000000002534. PMID 27673513